CLINICAL TRIAL: NCT05051384
Title: Using the Superb Microvascular Imaging Method in the Diagnosis of Intraocular Tumors (SMITIS)
Brief Title: Superb Microvascular Intraocular Tumor Imaging Study (SMITIS)
Acronym: SMITIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-AOIP-05; 2021-A01289-32 (Other: ANSM)
Record Dates: First submitted 2021-08-20; First posted 2021-09-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Ocular Tumor
MeSH Terms: conditions — Eye Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraocular tumor (Experimental): New sonographic software technique on ultrasonography to detect low-vascular flow inside intraocular tumors
  Interventions: Diagnostic Test: Doppler technology

INTERVENTIONS:
Diagnostic Test: Doppler technology — The study of tumor vascularization can help in the differential diagnosis and follow-up of tumors, and therefore can impact the management of patients with tumors

SUMMARY:
The diagnosis and monitoring of intraocular tumors are based on multimodal imaging in addition to the clinical examination (ultra-widefield retinal imaging, echography, angiography). Nevertheless, it may be difficult in cases of retinal hemorrhage, small tumor size or atypical presentation. The study of microvascular flow (Superb Microvascular Imaging, SMI) of intraocular tumors could improve the confidence of differential diagnosis when evaluating these suspicious lesions, or even determine whether a lesion is benign or malignant by describing the vascularization of the lesion.

The investigators propose to study the microvascular flow patterns of intraocular tumors prior to proton therapy.

DETAILED DESCRIPTION:
The ultrasound equipment available in ophthalmology does not have Doppler technology and does not allow the study of the vascularization and microvascularization of intraocular lesions. The interest in the system used in this study is to import SMI into ophthalmology to study tumor microvascularization. The study of tumor vascularization can help in the differential diagnosis and follow-up of tumors, and therefore can impact the management of patients with tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Intraocular tumor not previously treated with proton therapy

Exclusion Criteria:

* Severe active ocular, periocular or intraocular inflammation
* Intraocular pressure > 30 mmHg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
Qualitative description of the intratumoral microvascular flow | Visite 2 - two weeks after Day 0
  Number of visible feeding pedicles
Qualitative description of the intratumoral microvascular flow | Month 6
  Number of visible feeding pedicles

SECONDARY OUTCOMES:
quantification of microvascular flow for each tumor | Visite 2 2weeks after Day 0
  Presence or absence of arteriovenous shunts
quantification of microvascular flow for each tumor | month 6
  Presence or absence of arteriovenous shunts

CONTACTS AND LOCATIONS:
Overall Officials: Sacha NAHON ESTEVE, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France, France

IPD SHARING:
Plan to Share IPD: No